CLINICAL TRIAL: NCT04428541
Title: Determination of the Validity of a Questionnaire to Assess the Visual Function of Preverbal Children With Operable Bilateral Ocular Pathologies
Acronym: EVEIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PDU_2020_1
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Eye Diseases; Vision Disorders
Keywords: Eye Diseases; Vision Disorders; Questionnaire Design; Children; Infant
MeSH Terms: conditions — Eye Diseases; Vision Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire (Experimental): Description : 18 items questionnaire, filled by the parents of the child
  Interventions: Other: Questionnaire for visual function assessment of preverbal children

INTERVENTIONS:
Other: Questionnaire for visual function assessment of preverbal children — 18 items questionnaire

SUMMARY:
In some symmetrical pediatric ocular pathologies, the treatment is surgical with usually satisfactory postoperative results in visual terms.

However, it is often difficult to choose the right moment to operate. The main difficulty is that the child's vision is unknown since the child is still in a preverbal age.

The investigators have developed a questionnaire with the aim of quantifying the child's vision so that the decision is most justified. The items of this questionnaire were established based on the literature and were submitted to a panel of experts in ophthalmo-pediatrics. The objective of this study is to determine the internal validity and as far as possible (since there is no equivalent tool) the external validity of the questionnaire developed.

ELIGIBILITY:
Inclusion Criteria:

Common to the three groups:

* Patient aged 0 to 36 months
* Diagnosis of known ocular pathology

For patients targeted by the questionnaire:

- Patient with operable bilateral ocular pathology

For negative controls:

- Patient without ocular pathology inducing a decrease in vision

For positive controls:

* Patient with inoperable bilateral ocular pathology
* Patient without light perception

Exclusion Criteria:

* Patient with unilateral ocular pathology
* Verbal patients (able to express themselves through speech)

Ages: 0 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Measure the internal validity of the questionnaire developed to assess the visual acuity of preverbal children | Inclusion
  Reliability evaluated by Cronbach's alpha coefficient and its 95% confidence interval.
  unabbreviated scale title : Assessment of Visual Function in Preverbal Children in Bilateral Ocular Pathology
  Minimum value : 0
  Maximum value : 18
  Higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DUREAU, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A de Rothschild, Paris, France